CLINICAL TRIAL: NCT00182026
Title: A Randomized Trial of Diabetes Intervention in the Community to Help Achieve Reduced Glucose Elevation: Diabetes IN-CHARGE
Brief Title: Diabetes IN-CHARGE: Trial of Diabetes Intervention in the Community to Help Achieve Reduced Glucose Elevation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Hertzel Gerstein, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT-68786
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2009-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; community intervention; self-management; prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: personal feedback report — A computer-generated feedback report that provides personalized diabetes self-management recommendations to participants based on their responses to a self-administered questionnaire.

SUMMARY:
The purpose of this study is to test whether providing personalized diabetes self-management recommendations and feedback improves blood sugar control more than providing generalized diabetes educational material alone.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a common chronic disease that is rapidly rising in prevalence, affecting upwards of 35,000 adults in the Hamilton, Ontario region (population 400,000). The magnitude and growth of the problem and its serious health consequences suggest that:

1. diabetes is now a major public health problem; and
2. interventions at the community level are needed to mitigate its health impact.

During the last 5 years, Diabetes Hamilton was successfully piloted as a free community-based program available to anyone with diabetes. It promotes diabetes self-management, self-efficacy and awareness through the provision of generalized diabetes information (e.g. newsletters, workshops, forums, resource directories) to consumers, local physicians and other health professionals.

This trial will determine if supplementing Diabetes Hamilton with an automated tailored feedback system that:

1. provides information;
2. generates and communicates specific evidence-based recommendations to users from a self-administered questionnaire;
3. copies this communication to the patient's designated physician;
4. facilitates access to community resources; and
5. provides a simple way for the patient to track changes in indicators of health can improve A1c and other diabetes care indicators more than Diabetes Hamilton alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes of 1 or more years duration
* Health insurance coverage within Ontario
* Ages 40 or older
* Registered in, or willing to register in Diabetes Hamilton
* Able to read and understand English and provide informed consent in English
* Have home access to either mail, e-mail or the internet
* Have a baseline A1c >= 7%

Exclusion Criteria:

* Current pregnancy
* Residence in an institution that provides diabetes care
* Cohabiting with study participant
* Residence outside the city of Hamilton
* Inability to read or understand English
* Inability/unwillingness to sign the informed consent or comply with protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
A1c | 6 months and 1 year

SECONDARY OUTCOMES:
diabetes-related self-care behaviours, drug use, clinical outcomes | 6 months and 1 year
diabetes-specific quality of life | 1 year
incremental cost/quality-adjusted life-year [QALY] | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hertzel C Gerstein, MD MSc FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Sherifali D, Greb JL, Amirthavasar G, Hunt D, Haynes RB, Harper W, Holbrook A, Capes S, Goeree R, O'Reilly D, Pullenayegum E, Gerstein HC. Effect of computer-generated tailored feedback on glycemic control in people with diabetes in the community: a randomized controlled trial. Diabetes Care. 2011 Aug;34(8):1794-8. doi: 10.2337/dc11-0006. Epub 2011 Jun 16. PMID 21680723